CLINICAL TRIAL: NCT06748885
Title: Prospective, Multicentre, Non-randomised, Open Study Evaluating the Efficacy and Fixation of the Mpact 3D Metal Monolit Cup
Brief Title: Mpact 3D Metal Monolit Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.028.01
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Total Hip Arthroplasty (THA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mpact 3D Metal Monolith — THA with Mpact 3D Metal Monolith

SUMMARY:
Total hip arthroplasty (THA) is one of the most common operations performed in orthopaedics to improve a patient's quality of life.

Surgeons are constantly seeking to improve all aspects of care related to this procedure, whether it be improving implant technology, improving instrumentation or the technique involved in performing the procedure.

In recent years, a new porous titanium coating has been introduced to promote good osseointegration of uncemented cups. High friction torque and a feeling of immediate anchorage provide excellent primary stability, while high porosity ensures bone growth providing secondary stability. With higher porosity than standard coatings, a greater volume of bone can be present in the porous surface, giving a proportional increase in force at the interface. he Mpact 3D Metal Monolith cup has been designed to provide greater range of motion and improved joint stability, with a reduced risk of dislocation. It is an innovative design that improves stability and provides a favourable environment for long-term biological metal-bone fixation.

The current study aims to collect clinical and radiological data to assess the function of the operated hip and the stability of the Mpact 3D Metal Monolith cup at 2 years and survival at 5 years for the treatment of patients requiring hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a disease that corresponds to the indications for use of Medacta implants (according to the instructions for use)
2. Patient eligible for primary total hip arthroplasty
3. Patient aged between 18 and 75 years
4. Patient covered by the French Social Security system or an equivalent protection scheme.
5. Patient able, in the investigator's opinion, to comply with the requirements of the study.

Exclusion Criteria:

1. Patient suffering from inflammatory arthritis
2. Previously operated hip
3. Patient requiring a transplant
4. Hip tumour involved
5. Patient with progressive local or systemic infection
6. Severe acetabular dysplasia
7. Patient with muscle loss, neuromuscular disease or vascular impairment of the affected limb.

4. Patient with known medical problems that may compromise independent recovery of mobility 5. Patient with a BMI greater than 40 kg/m². 6. Patient with major cognitive impairment that prevents him/her from fully understanding the requirements of the study 7. Patient living in a geographical area where study follow-up is not possible. 8. Patient taking part in interventional research 9. Minor patient 10. Protected adult patient 11. Vulnerable person according to article L1121-6 of the Public Health Code

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the hip function | Preoperative, 3 months, 6 months, 1 year, 2 years, 5 years
  The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The original version was published 1969[1]. The HHS is an outcome measure administered by a qualified health care professional, such as a physician or a physical therapist. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

SECONDARY OUTCOMES:
Analysis of the primary stability of the implant at 2 years | 2 years
  Protocol EBRA-Cup: Measurement of longitudinal/transversal migration of acetabular cup in digital serial radiographs (minimum of 4 x-rays per series). Full size AP pelvis radiographs are required.
  Accuracy: +/- 1mm.
Analysis of the wear of the polyethylene insert (HighCross) at 2 years | 2 years
  Martell method of linear wear measurement
Evaluation of the fixation and osteolysis | Immediate postoperative, 3 months, 6 months, 1 year, 2 years, 5 years
  Radiological analysis
Evaluation of the mobility | Preoperative, 3 months, 6 months, 1 year, 2 years, 5 years
  The Oxford Hip Score (OHS) is a joint-specific, patient-reported outcome measure designed to assess disability in patients undergoing total hip replacement. The OHS is a short 12-item survey that can be done with pen and paper. Patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains (pain and function) with six items or questions in each. Each item has five possible responses. In the original scoring responses were from 1 = least difficult to 5= most difficult. Item scores are summed to give a total score from anywhere between 12 and 60. The lower the score, the better the outcome.
Evaluation of the safety of the implant | Intraoperative, immediate postoperative, 3 months, 6 months, 1 year, 2 years, 5 years
  Collection of intraoperative and postoperative complications
Evaluation of the survival of the implant | 3 months, 6 months, 1 year, 2 years, 5 years
  Kaplan-Meier survival method

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique Brétéché, Nantes
  - Hôpital Lariboisière, Paris
  - Hôpital Cochin, Paris